CLINICAL TRIAL: NCT03285464
Title: Investigating the Effects of a Triplanar Rotary Based Hip Focused Therapeutic Exercise Program on Dynamic Lower Extremity Alignment and Functional Performance
Brief Title: Utilizing the Trunk as a Proximal Lever to Strengthen the Hip Musculature and Alter Lower Extremity Function
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: High Point University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 201508-387
Record Dates: First submitted 2017-09-12; First posted 2017-09-18 (Actual); Last update posted 2018-02-26 (Actual); Status verified 2018-02

CONDITIONS: Patellofemoral Pain Syndrome
Keywords: knee; hip; exercise; proximal control; PFPS
MeSH Terms: conditions — Patellofemoral Pain Syndrome; Motor Activity

STUDY DESIGN:
Intervention Model Description: One group will do current hip focused intervention published previously second group will receive a new hip intervention and then pre/post testing will take place for static and dynamic kinematics and hip strength
Who Masked: Participant
Masking Description: Only the subjects will not know which group they are being assigned to
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Hip (Active Comparator): This group will perform a known hip strengthening program
  Interventions: Other: Triplanar Rotary Resistance
- Trunk (Experimental): This group will use the trunk as a lever to strengthen the hip
  Interventions: Other: Triplanar Rotary Resistance

INTERVENTIONS:
Other: Triplanar Rotary Resistance — Trunk group will strengthen the hip using the trunk as a lever to access the hip. The hip group will use femur as the lever to strengthen the hip.
  Other Names: Convention Hip Focused

SUMMARY:
Does a rotary based triplanar exercise intervention that utilizes the trunk as a proximal lever, strengthen the hip and alter dynamic LE alignment in running females?

DETAILED DESCRIPTION:
Current hip-focused programs fail to alter hip adduction angles in females while performing higher speed and more complex maneuvers such as running.

(Willy, et al., 2011) - 10 female runners, underwent 6 wk. hip focused intervention, change in SLS but NO change in hip adduction angle while running.

A different intervention strategy that includes utilizing the trunk as the proximal lever to strengthen the hip, could potentially alter biomechanical outcomes such as hip adduction angles in female runners.

This study will apply a new intervention model and then measure running, single leg squat and hip strength to determine if a newly informed intervention can alter LE kinematics in females while running and make improvements in hip strength following the intervention Inclusion Criteria

* 18 years old or greater
* Female Exclusion Criteria
* Injury of the lumbar spine, hips, knees or foot/ankle in the last 6mos that required medical attention
* any surgery of the lower back or the pelvis or lower extremities any time in the subjects life

ELIGIBILITY:
Inclusion Criteria:

* 18> year old female; must be able to run on the treadmill for 5-7 min and perform a single leg squat

Exclusion Criteria:

* surgery to the LB or lower extremities Significant injury (seeking medical attention) to the LB or LEs in the last 6mos.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Include only females
Enrollment: 32 (Actual)
Dates: Start 2017-08-09 (Actual); Primary Completion 2017-12-15 (Actual); Study Completion 2017-12-15 (Actual)

PRIMARY OUTCOMES:
Change in Hip Strength after a 12 week hip focused intervention | Baseline measures at initial data collection; repeat post intervention measures at 6wks
  Isometric hand held dynamometer

SECONDARY OUTCOMES:
Biomechanical assessment of single leg squat | Baseline measures at initial data collection; repeat post intervention measures at 6wks
  Subject squats on single leg and qualitative scoring is administered to determine the subjective amount of contralateral pelvic drop and femoral adduction to be described as dynamic knee valgus. The qualitative values will be binary in nature, whereas DKV is present or not.
Biomechanical Running Assessment | Baseline measures at initial data collection; repeat post intervention measures at 6wks
  2/3D analysis of running gait following intervention; Utilizing both 3D/2D methods the measure of contralateral pelvic drop and the bisection of the patella will determine the amount of femoral adduction noted during running. The change in the femoral adduction angle after a 6 week intervention is the specific outcome measure to be obtained.

CONTACTS AND LOCATIONS:
Overall Officials: Alexis Wright, DPT, Principal Investigator — HPU; Eric Hegedus, DPT, Study Chair — HPU; Kevin Ford, PhD, Study Director — HPU
Locations (1):
- High Point University, High Point, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Undecided
The data collected will only be shared amongst the research team named in this protocol.